CLINICAL TRIAL: NCT04539301
Title: Multicentric Prospective Validation of a Universal Test to Quantify Apixaban, Rivaroxaban, Danaparoid and Fondaparinux Levels
Acronym: UniXa
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0061
Record Dates: First submitted 2020-09-01; First posted 2020-09-04 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Anticoagulation; Venous Thromboembolism; Atrial Fibrillation
Keywords: Anticoagulants (MeSH); Blood Coagulation Tests (MeSH); Drug monitoring (MeSH); Factor Xa Inhibitors (MeSH); Heparin (MeSH)
MeSH Terms: conditions — Venous Thromboembolism; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation cohort: In the derivation cohort, we will determined the conversion factor linking apixaban, rivaroxaban, fondaparinux, or danaparoid measured level, on the one hand, and heparin anti-Xa activity, on the other hand.
  Interventions: Diagnostic Test: Estimated anticoagulant level (conversion factor x anti-Xa activity)
- Validation cohort: In the validation cohort, for each tested anticoagulant, we will used the conversion factor determined in the derivation cohort to infer the estimated level of anticoagulant from heparin anti-Xa activity:
  estimated anticoagulant level = conversion factor for this anticoagulant × heparin anti-Xa activity
  The agreement between measured and estimated levels of each factor-Xa inhibitor will be assessed.
  Interventions: Diagnostic Test: Estimated anticoagulant level (conversion factor x anti-Xa activity)

INTERVENTIONS:
Diagnostic Test: Estimated anticoagulant level (conversion factor x anti-Xa activity) — Estimated anticoagulant level (conversion factor x anti-Xa activity)

SUMMARY:
Despite their usefulness in perioperative and acute care settings, factor-Xa inhibitors-specific assays are scarcely available, contrary to heparin anti-Xa assay. The investigators aimed at assessing whether the widely used heparin anti-Xa assay can quantify the apixaban, rivaroxaban, fondaparinux and danaparoid levels.

ELIGIBILITY:
Inclusion Criteria :

* Blood sample from adult patients treated with apixaban or rivaroxaban or danaparoid or fondaparinux

Exclusion Criteria :

* Patients treated with unfractionated heparin or low molecular weight heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated with apixaban or rivaroxaban or danaparoid or fondaparinux
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Agreement between measured and estimated levels of each factor-Xa inhibitor | 2 years
  An estimated anticoagulant level between 80 and 120% of the value obtained by the reference method ("specific assay") will be deemed clinically acceptable, i.e. the patient's management would have been the same.

SECONDARY OUTCOMES:
Evaluation of the performance of the estimated anticoagulant level method by an inter-laboratory comparison program | 2 years
Cost comparison (estimated anticoagulant level method versus specific dosage) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No